CLINICAL TRIAL: NCT00310934
Title: Graded Strategy for Pharmacological Treatment of Heroin Dependence
Brief Title: A Stepwise Strategy Utilizing Buprenorphine and Methadone
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Collaborators: Swedish National Drug Policy Coordinator (Unknown); Region Stockholm (Other Government); Schering-Plough (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KarolinskaUH Regional 373/03
Record Dates: First submitted 2006-04-03; First posted 2006-04-05 (Estimated); Last update posted 2006-10-24 (Estimated); Status verified 2006-03

CONDITIONS: Heroin Dependence
Keywords: heroin dependence; methadone; buprenorphine; contingency management; relapse prevention
MeSH Terms: conditions — Heroin Dependence | interventions — Methadone; Buprenorphine; Secondary Prevention

INTERVENTIONS:
Drug: methadone
Drug: buprenorphine / methadone sequence
Behavioral: Relapse prevention
Behavioral: Contingency management

SUMMARY:
The objective of this study is to compare optimally given methadone maintenance treatment (MMT) for heroin dependence with a novel, sequential strategy, where patients are offered buprenorphine as first line treatment, allowed dose adjustments as needed, and switched to methadone if the maximal dose of buprenorphine is insufficient.

DETAILED DESCRIPTION:
The objective of this study is to compare optimally given methadone maintenance treatment (MMT) for heroin dependence with a novel, sequential strategy (STEP), where patients are offered buprenorphine as first line treatment, allowed dose adjustments as needed, and switched to methadone if the maximal dose of buprenorphine is insufficient.

For this purpose, 96 subjects at two centers (Uppsala and Stockholm) are randomized to MMT or STEP and followed for 6 months. Retention in treatment is the primary outcome. Secondary outcomes in completers are proportion urine samples free of illicit opiates on app. twice weekly sampling, and problem severity as measured by a semistructured interview, the Addiction Severity Index (ASI) at baseline and after 3 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Heroin dependence according to DSM IV > 1year
* Age > 20 years
* Acceptance of the stated treatment principles.

Exclusion Criteria:

* Severe psychiatric illness such as dementia or psychosis compromising the patient's ability to provide informed consent
* Other clinically significant psychiatric illness unless stable under treatment
* Severe medical condition such as advanced lung disease, unstable cardiovascular disease, severe liver disease
* Other clinically significant medical condition unless stable under treatment
* Treatment with anti-seizure drugs or disulfiram
* Pregnancy or intent to become pregnant within the next year
* Ongoing nursing
* Patients involuntarily discharged from a methadone or buprenorphine maintenance program within the last 3 months not eligible.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96
Dates: Start 2005-08; Study Completion 2006-03

PRIMARY OUTCOMES:
Retention in treatment

SECONDARY OUTCOMES:
Proportion urine samples free of illicit drugs
Problem severity as measured by Addiction Severity Index

CONTACTS AND LOCATIONS:
Overall Officials: Markus Heilig, MD PhD, Principal Investigator — Karolinska Institute, Stockholm
Locations (1):
- Dept of Clinical Neuroscience, Karolinska Inst, Stockholm, Sweden